CLINICAL TRIAL: NCT01260207
Title: Using Interactive Voice Response to Improve Disease Management and Compliance With Acute Coronary Syndrome Best Practice Guidelines
Brief Title: Using IVR to Maintain ACS Patients on Best Practice Guidelines
Acronym: IVR-ACS BPG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to unachievable sample size and lack of resource availability
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-07-391
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-03

CONDITIONS: Acute Coronary Syndrome; Medication Adherence
Keywords: Acute Coronary Syndrome; Interactive Voice Response Technology; Best Practice Guidelines; Compliance; Health Care Utilization
MeSH Terms: conditions — Acute Coronary Syndrome; Medication Adherence; Patient Compliance; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVR group (Experimental): Patients in this arm will receive IVR follow-up telephone calls at 1,3,6,9 and 12 months post-discharge consisting of predetermined questions related to medication management, smoking cessation, diet, exercise and education as recommended by the ACC/AHA BPG for ACS. Upon completion of the IVR follow-up, all patients will be called by a member of the clinical research staff and asked to complete a follow-up survey.
  Interventions: Other: IVR group
- Usual care (No Intervention): Patients in this arm will not receive IVR follow-up. One year after discharge, all patients will be called by a member of the clinical research staff and asked to complete a follow-up survey.

INTERVENTIONS:
Other: IVR group — Patients in this arm will receive IVR follow-up telephone calls at 1,3,6,9 and 12 months post-discharge consisting of predetermined questions related to medication management, smoking cessation, diet, exercise and education as recommended by the ACC/AHA BPG for ACS. Upon completion of the IVR follow-up, all patients will be called by a member of the clinical research staff and asked to complete a follow-up survey.
  Other Names: Assignment to Interactive Voice Response
  Arms: IVR group

SUMMARY:
The purpose of this study is to determine whether interactive voice response (IVR) technology can be used to bring post discharge care for acute coronary syndrome (ACS) closer to best practice guidelines (BPGs).

The study hypothesis is that ACS patients who are contacted by IVR technology will be more likely to receive care as recommended in the BPGs than those followed by usual care.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is a significant public-health problem in Canada and worldwide with 20,000 Canadians dying of myocardial infarction and 42,000 dying of coronary artery disease in 1999. Large clinical trials have provided evidence for the development of standardized best practice guidelines (BPG) and compliance with these guidelines have significantly improved survival. Despite the development and dissemination of BPG, their application in patients with ACS is suboptimal. This randomized control trial will use 2 groups: IVR and usual care. Patients in the IVR group will receive 5 automated calls at 1,3,6,9 and 12 months consisting of predetermined questions related to medication management, smoking cessation, diet, exercise and education as recommended by the ACC/AHA BPG for ACS. Responses are captured in a database allowing for interventions to maintain patients on BPG as needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from LHSC with ACS (acute myocardial infarction, STEMI, NSTEMI or unstable angina)
* Patients who have a land line telephone service at home
* Patients who speak English

Exclusion Criteria:

* Patients discharged to a care facility or transferred to another health care institution
* Patients who cannot provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-12-15 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
Compliance with BPGs | 1 Year

SECONDARY OUTCOMES:
Utilization of health care resources: emergency visits, unscheduled physician visits and hospitalization and patient satisfaction | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Neville G. Suskin, MBChB, MSc, Principal Investigator — University of Western Ontario and London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada